CLINICAL TRIAL: NCT02449746
Title: An Unblinded Study of the Feasibility of Plasmapheresis or Intravenous Immunoglobulin, Combined With Corticosteroids, in Patients With Acute Psychosis Associated With Anti-neuronal Membrane Auto-antibodies
Brief Title: Study of Immunotherapy in Autoantibody Positive Psychosis
Acronym: SINAPPS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Oxford (Other); Stanley Medical Research Institute (Other); McPin Foundation (Other)
Responsible Party: Principal Investigator, Alasdair Coles, Prof Rev Alasdair Coles, Principal Investigator, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 609/M/C/1368
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia; Psychosis; Auto Immune Disorders
Keywords: Schizophrenia; Psychosis; Mental Health; Autoimmunity; Psychoneuroimmunology
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Psychological Well-Being; Autoimmune Diseases | interventions — Plasma Exchange; Immunoglobulins, Intravenous

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Immunoglobulin (IVIG) (Active Comparator): Intravenous Immunoglobulin IVIG is a pooled blood product from 3000-100,000 human blood donors with direct immunomodulatory effects.
  IVIG will be given at a dose of 2g/kg over 4 days. Dosing at 2g/kg is established in neurological disorders, with limited evidence that lower doses are less effective although adequate dosing studies have not been performed.
  Interventions: Biological: Intravenous immunoglobulin
- Plasma Pheresis / Plasma Exchange (PLEX) (Active Comparator): Plasma Exchange (PLEX) is a procedure in which the subject's blood is passed through a medical device which separates out plasma from the other blood components, and replaces the plasma with albumin or plasma or other colloid. PLEX therefore removes circulating pathogenic antibodies, and its use was first reported in myasthenia gravis in 1976, and furthermore therapeutic benefit after PLEX supports an antibody mediated pathogenesis of disease. In PLEX, 200-250 mL plasma per kg body weight is exchanged typically over 7-14 days using 5% albumin as replacement, often at alternate days which increases the amount of immunoglobulin removed due to equilibrium effects . PLEX modality (centrifugation or filtration), type of anticoagulation, and dose scheduling will be determined by local centre practice
  Interventions: Biological: Plasma Exchange

INTERVENTIONS:
Biological: Plasma Exchange — PLEX is a procedure in which the subject's blood is passed through a medical device which separates out plasma from the other blood components, and replaces the plasma with albumin or plasma or other colloid. PLEX therefore removes circulating pathogenic antibodies, and furthermore therapeutic benefit after PLEX supports an antibody mediated pathogenesis of disease. In PLEX, 200-250 mL plasma per kg body weight is exchanged typically over 7-14 days using 5% albumin as replacement, often at alternate days which increases the amount of immunoglobulin removed due to equilibrium effects. PLEX modality (centrifugation or filtration), type of anticoagulation, and dose scheduling will be determined by local centre practice.
  Other Names: PLEX
  Arms: Plasma Pheresis / Plasma Exchange (PLEX)
Biological: Intravenous immunoglobulin — Active Comparator: Intravenous Immunoglobulin (IVIG) IVIG is a pooled blood product from 3000-100,000 human blood donors with direct immunomodulatory effects.
  IVIG will be given at a dose of 2g/kg over 4 days. Dosing at 2g/kg is established in neurological disorders, with limited evidence that lower doses are less effective although adequate dosing studies have not been performed.
  Other Names: IVIG
  Arms: Intravenous Immunoglobulin (IVIG)

SUMMARY:
Psychosis is a mental health problem that causes people to perceive or interpret things differently from those around them, often involving hallucinations or delusions. Psychosis and schizophrenia are common disorders which predominantly affect younger adults. Recently, the investigators discovered that 5-10% of people with psychosis have antibodies in the blood that are capable of targeting the surface of brain cells, specific to the N-methyl-D-aspartate (NMDA) receptor or voltage gated potassium channel complex, which the investigators believe may be causing the problem. Those positive for antibodies may have a problem with their immune system and this may prevent their brain from working normally. This trial aims to test the feasibility of removing or reducing the antibodies in patients' blood, using immunotherapy, and see if this improves symptoms of psychosis. Immunotherapy in this feasibility study will involve giving all patients steroid tablets and half of them will also receive a drug called "intravenous immunoglobulin" whereas the other half will have a procedure called "plasma exchange". The feasibility study is designed to identify which method of immunotherapy is most suitable for use in this patient population.

Results from this will inform on the methodology used for a proposed larger randomised control trial.

DETAILED DESCRIPTION:
An autoimmune disease occurs when a person's immune system begins to respond to normal bodily substances and tissues as if it were foreign or related to disease. There are a number of autoimmune disorders, some of which can affect the brain by targeting the surface of brain cells, for example signalling proteins like the NMDA receptor or voltage gated potassium channel complex. Some cases of encephalitis, a disorder of brain inflammation that can be autoimmune, are caused by these antibodies, but often present with psychotic experiences, such as hallucinations, and may see a psychiatrist at this stage, before they go on to experience seizures and brain swelling, and are seen by a neurologist. These patients are treated with immunotherapy, and after treatment see a reduction in both seizures and psychotic symptoms.

Recently the investigators identified patients with psychosis who test positive for these antibodies, but do not go on to experience these other symptoms of encephalitis. It has been suggested that these patients suffer from an autoimmune disorder similar to the encephalitis described above. Small pilot studies in these antibody positive psychosis patients have shown various immunotherapies can reduce both symptoms of psychosis and number of autoantibodies present in their blood. A randomised clinical trial (RCT) is required to confirm this. However a feasibility study is required first to investigate whether it is possible to deliver the immunotherapy treatments in patients with psychosis. The treatments require an infusion over a few hours (IVIG) or an admission to an acute medical ward for several days(plasma exchange). Both may be challenging for people who are paranoid or agitated. The investigators need to assess whether it is possible to deliver these treatments before proceeding to a large scale, clinical trial.

This is a multicentre, randomised, uncontrolled, open label feasibility study. Patients with psychosis and a positive blood test for antibodies will be identified from one of 24 recruiting centres across England. They will undergo screening assessment for eligibility (interview with psychiatrist and neurologist and baseline investigations where possible, including MRI, EEG and lumbar puncture) and give informed consent for the study. A further blood sample (10ml) will be taken for future research. 10 Participants will be randomised to one of two clinical care pathways: either an infusion of intravenous immunoglobulins, or plasma exchange treatment. Both groups will receive steroid tablets, and both groups will continue to receive psychiatric treatment, including antipsychotic medication, as normal.

At two months after randomisation the research team will speak to the treating clinicians to gather the primary outcome measure which is whether the patient received the allocated treatment within two weeks of allocation. The researchers may also confirm this outcome from the clinical records.

ELIGIBILITY:
Inclusion Criteria:

* Acute psychosis
* Serum and/or Cerebrospinal flud (CSF) neuronal membrane autoantibodies (including N-methyl-D-aspartate receptor (NMDAR), Voltage gated potassium channel (VGKC), Leucine-rich, glioma inactivated 1,(LGI1), gamma-aminobutyric acid (GABA [A]) receptor)
* Positive and Negative Syndrome Scale (PANSS) >4 on items of positive psychotic symptoms

Exclusion Criteria:

* current symptoms greater than 2 years duration,
* co-existing severe neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who start on allocated care pathway within 2 weeks of randomisation. | 2 weeks
  percentage of recruited patients who start on allocated care pathway within 2 week from randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Coles, 01223 762016, Principal Investigator — ajc1020@medschl.cam.ac.uk
Locations (5):
- United Kingdom (5):
  - University Hospitals Birmingham, Birmingham
  - Cambridge University Hospitals, Cambridge
  - Nottingham University Hospitals, Nottingham
  - Oxford University Hospitals, Oxford
  - University Hospitals Southampton, Southampton